CLINICAL TRIAL: NCT07366125
Title: THE EFFECT OF SCENARİO-BASED SİMULATİON METHOD ON NURSİNG STUDENTS' BASİC LİFE SUPPORT PRACTİCE SKİLLS AND SELF-EFFİCACY LEVELS: A CONTROLLED EXPERİMENTAL STUDY
Brief Title: EFFECT OF SCENARIO-BASED SIMULATION ON BASIC LIFE SUPPORT SKILLS AND SELF-EFFICACY IN NURSING STUDENTS
Acronym: SBS-BLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Ekrem EKER, Registered Nurse, MSc Student, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BARUN-MSC-TYD-01
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Basic Life Support Training
Keywords: Nursing; scenario; simulation; student; basic life support; practical skills; self-efficacy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group or the control group. The intervention group received scenario-based simulation training, while the control group received standard basic life support training. Both groups were followed in parallel throughout the study period.
Masking Description: No blinding was applied in this study; both participants and researchers were aware of the group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Scenario-Based Simulation Group (Experimental): Participants in this group received scenario-based simulation training on basic life support.
  Interventions: Other: Scenario-Based Simulation Training
- Arm 2: Standard Training Group (Active Comparator): Participants in this group received standard theoretical and practical training on basic life support according to the nursing curriculum.
  Interventions: Other: Standard Basic Life Support Training

INTERVENTIONS:
Other: Scenario-Based Simulation Training — Scenario-based simulation training was provided to improve basic life support skills and self-efficacy among nursing students.
  Other Names: Simülasyon Tabanlı Temel Yaşam Desteği Eğitimi
  Arms: Arm 1: Scenario-Based Simulation Group
Other: Standard Basic Life Support Training — Hemşirelik müfredatına uygun olarak verilen standart teorik ve pratik temel yaşam desteği eğitimi.
  Arms: Arm 2: Standard Training Group

SUMMARY:
This study aimed to evaluate the effectiveness of scenario-based simulation in improving nursing students' adult basic life support (ABLS) skills and self-efficacy. Ethical approval was obtained from the Bartın University Social and Human Sciences Ethics Committee, and institutional permission was granted. The study was conducted with students from the Department of Nursing at the Faculty of Health Sciences, Bartın University, between October and December 2025.

The sample size was determined based on the literature using an alpha level of 0.05, an effect size of 0.63, and a statistical power of 85%. A total of 50 students who met the inclusion criteria were randomly assigned to either the experimental or control group. All participants were informed about the study and provided written informed consent.

Data were collected using the Student Information Form, the Adult Basic Life Support Knowledge Level Assessment, the Adult Basic Life Support Skill Performance Assessment Form, and the Student Self-Efficacy Scale. All students received a 90-minute theoretical ABLS training delivered by an experienced researcher. Following the theoretical session, the control group practiced ABLS using the demonstration method on a feedback-enabled manikin, while the experimental group practiced using scenario-based simulation. Both applications were conducted under academic supervision.

Students' knowledge, skill performance, and self-efficacy levels were assessed immediately after training, after the first application, and at a one-month follow-up. Data were analyzed using SPSS version 29.0. No significant difference was found between the groups in knowledge scores immediately after training. After the first application, no significant differences were observed in knowledge or self-efficacy levels; however, skill performance scores were significantly higher in the control group. At the one-month follow-up, a significant decline in skill performance was observed in the control group, whereas the experimental group maintained their performance levels.

These findings indicate that scenario-based simulation supports the long-term retention of practical ABLS skills. Therefore, integrating simulation-based methods into adult basic life support education in nursing programs is recommended.

DETAILED DESCRIPTION:
This study aimed to examine the effectiveness of scenario-based simulation methods in improving nursing students' adult basic life support skills and self-efficacy levels. Ethical approval was obtained from the Bartın University Social and Human Sciences Ethics Committee, and official permission was granted by the relevant institution. The study was conducted with students from the Department of Nursing at the Faculty of Health Sciences, Bartın University. Data were collected between October and December 2025. The sample size was calculated based on the literature with an alpha level of 0.05, an effect size of 0.63, and a statistical power of 85 percent. The study was completed with 50 students who met the inclusion criteria and were randomly assigned to either the experimental group or the control group. All participants were informed about the research process, and their voluntary informed consent was obtained. Data were collected using the Student Information Form, the Adult Basic Life Support Knowledge Level Assessment, the Adult Basic Life Support Skill Performance Assessment Form, and the Student Self-Efficacy Scale. All students received a 90-minute theoretical adult basic life support training provided by a researcher with professional experience in the field. Following the theoretical training, students in the control group performed adult basic life support practices using the demonstration method on a feedback-enabled training manikin under academic supervision. Students in the experimental group performed adult basic life support practices using scenario-based simulation under the same supervision. Students' knowledge levels, skill performance, and self-efficacy levels were evaluated immediately after the training, during the first application, and at a one-month follow-up. Data analysis was performed using SPSS version 29.0. The findings indicated no significant difference between the groups in knowledge scores immediately after training. While no significant differences were observed in knowledge and self-efficacy levels after the first application, skill performance scores were significantly higher in the control group. However, at the one-month follow-up, a significant decline in skill performance was observed in the control group, whereas no significant decrease was found in the experimental group. These results suggest that scenario-based simulation provides a more sustainable improvement in practical skill performance. Therefore, it is recommended that adult basic life support education in nursing programs be supported with simulation-based methods.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in all stages of the research (pre-test - training - post-test, etc.),
* Actively enrolled in a Nursing Undergraduate Program,
* Able to read and understand Turkish,
* Not having any physical or cognitive disability that would prevent participation in practical training,
* Not having received any prior training in TYD (Basic Nursing Education).

Exclusion Criteria:

* Having received any non-research-related training on TYD that you can conduct research on previously,
* Being a graduate of a Health Vocational High School or a graduate of any associate's or bachelor's degree program in the health field,
* Not having registered for courses in the relevant period or having suspended the semester,
* Not regularly attending training sessions during the research process,
* Having serious health problems that will increase the data collection period,
* Incomplete completion of pre-test or post-test forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Basic Life Support Practice Skills | Baseline (pre-test), immediately after the intervention (post-test), and 1-month follow-up
  Basic life support practice skills were assessed using a standardized skills performance checklist.

CONTACTS AND LOCATIONS:
Overall Officials: EKER, Principal Investigator — Bartin University Faculty of Health Sciences
Locations (1):
- Bartin University Faculty of Health Sciences, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.